CLINICAL TRIAL: NCT01523587
Title: LUX-Lung 8: A Randomized, Open-label Phase III Trial of Afatinib Versus Erlotinib in Patients With Advanced Squamous Cell Carcinoma of the Lung as Second-line Therapy Following First-line Platinum-based Chemotherapy
Brief Title: LUX-Lung 8: A Phase III Trial of Afatinib (BIBW 2992) Versus Erlotinib for the Treatment of Squamous Cell Lung Cancer After at Least One Prior Platinum Based Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.125; 2011-002380-24 (EudraCT Number)
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Erlotinib Hydrochloride

ARMS (2):
- Afatinib (Experimental): Patients receive afatinib tablets once daily
  Interventions: Drug: afatinib
- Erlotinib (Active Comparator): Patients receive erlotinib tablets once daily
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: afatinib — Afatinib taken once daily, continuously until disease progression or unacceptable toxicity.
  Arms: Afatinib
Drug: erlotinib — erlotinib taken once daily
  Arms: Erlotinib

SUMMARY:
This randomised, open-label phase III trial will be performed in patients with advanced squamous cell carcinoma of the lung requiring second-line treatment after receiving first-line platinum-based chemotherapy. The primary objective of this trial is to compare the efficacy of BIBW 2992 to erlotinib as second-line treatment in this group of patients.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of advanced stage NSCLC squamous histology.
2. Platinum-based doublet chemotherapy as 1st line treatment of Stage IIIB/IV NSCLC.
3. Eligible to receive 2nd line therapy in the opinion of the investigator.
4. Measurable disease according to RECIST 1.1.
5. Adequate Performance Status.
6. Availability of tumour tissue material for correlative studies. Archived tumour tissue is acceptable.
7. Adequate organ function.
8. Age = 18 years and above.
9. Written informed consent that is consistent with International Conference on Harmonisation (ICH)-Good Clinical Practice (GCP) guidelines.

Exclusion criteria:

1. Prior treatment with Epidermal Growth Factor Receptor (EGFR) directed small molecules or antibodies.
2. Radiotherapy within 4 weeks prior to randomization.
3. Active brain metastases .
4. Any other current malignancy or malignancy diagnosed within the past three (3) years (other than basal-cell carcinoma of the skin, in situ cervical cancer, in situ prostate cancer).
5. Known pre-existing interstitial lung disease.
6. Significant or recent acute gastrointestinal disorders with diarrhoea as a major symptom
7. Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
8. Women of child-bearing potential and men who are able to father a child, unwilling to be abstinent or use adequate contraception prior to study entry, for the duration of study participation and for at least 2 months after treatment has ended.
9. Female patients of childbearing potential (see Section 4.2.3.3) who:

   1. are nursing or
   2. are pregnant or
   3. are not using an acceptable method of birth control, or do not plan to continue using this method throughout the study and/or do not agree to submit to pregnancy testing required by this protocol.
10. Active hepatitis B infection (defined as presence of Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier.
11. Known or suspected active drug or alcohol abuse in the opinion of the investigator.
12. Any contraindications for therapy with afatinib or erlotinib.
13. Known hypersensitivity to erlotinib, afatinib or the excipients of any of the trial drugs.
14. Major surgery within 4 weeks of starting study treatment.
15. Prior participation in an afatinib clinical study, even if not assigned to afatinib.
16. Use of any investigational drug within 4 weeks of randomisation (unless a longer time period is required by local regulations or by the guidelines for the investigational product).
17. Patients without Progression of their lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2012-03-05 (Actual); Primary Completion 2013-10-21 (Actual); Study Completion 2017-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (191):
- United States (32):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - University of California, La Jolla, California
  - Sutter Medical Group, Sacramento, California
  - Boca Raton Reginl Hospital-Lynn Cancer Institute, Boca Raton, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Cancer Care of North Florida, PA, Lake City, Florida
  - Illinois Cancer Specialists, Niles, Illinois
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - University of Louisville, Louisville, Kentucky
  - West Jefferson General Hospital and Cancer Clinic, Marrero, Louisiana
  - Lahey Clinic, Burlington, Massachusetts
  - Commonwealth Hematology-Oncology, PC, Lawrence, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Queens Medical Associates, Fresh Meadows, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Mid Ohio Oncology/Hematology, Inc, Columbus, Ohio
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oncology Hematology Associates of Norhtern Pennsylvania, PC, DuBois, Pennsylvania
  - Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Temple University Cancer Center, Philadelphia, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Center of Cookeville Regional Medical Center, Cookeville, Tennessee
  - Paris Cancer Center (PCC), Texas Oncology, Paris, Texas
  - Cancer Therapy and Research at UTHSCSA, San Antonio, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Blue Ridge Cancer Care, Christiansburg, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Argentina (5):
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma de Bs As
  - Instituto Oncologico de Cordoba, Córdoba
  - Clínica Colombo S.A., Córdoba
  - Centro Oncologico de Rosario, Rosario
  - Centro Oncologico CAIPO, San Miguel de Tucumán
- Austria (4):
  - Medical University of Innsbruck, Innsbruck
  - LKH Leoben, Leoben
  - AKH d. Stadt Linz, Pulmologie, Linz
  - SMZ Baumgartner Hoehe Otto Wagner Spital, Vienna
- Canada (5):
  - BC Cancer Agency - Fraser Valley Centre, Surrey, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
- Chile (4):
  - Centro Oncologico Antofagasta, Antofagasta
  - Instituto de Terapias Oncologicas Providencia, Providencia, Santiago
  - Centro Internacional de Estudios Clinicos - CIEC, Recoleta, Santiago de Chile
  - Orlandi Oncologia, Vitacura
- China (9):
  - Beijing Cancer Hospital, Beijing
  - Beijing Hospital, Beijing
  - First Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central South University, Changsha
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - the 81th Hospital of PLA, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
- Denmark (3):
  - Herlev Hospital, Herlev
  - Næstved Sygehus, Næstved
  - Odense Universitetshospital, Odense C
- France (20):
  - HOP d'Angers, Angers
  - INS Bergonié, Bordeaux
  - HOP Côte de Nacre, Caen
  - HOP de Chauny, Chauny
  - HOP Gabriel-Montpied, Clermont-Ferrand
  - HOP de Creteil, Pneumo, Creteil, Créteil
  - HOP Le Mans, Le Mans
  - CTR Oscar Lambret, Cancéro, Lille, Lille
  - HOP Calmette, Lille
  - INS Paoli-Calmettes, Marseille
  - HOP Nord, Marseille
  - HOP de Mulhouse, Onco, Mulhouse, Mulhouse
  - HOP Cochin, Paris
  - HOP Val de Grâce, Onco, Paris, Paris
  - INS Jean Godinot, Onco, Reims, Reims
  - HOP de Rennes, Pneumo, Rennes, Rennes
  - HOP Saint Quentin, Onco, Saint Quentin, Saint-Quentin
  - HOP Civil, Strasbourg
  - HOP Foch, Suresnes
  - INS Gustave Roussy, Villejuif
- Germany (10):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Lungenklinik Hemer, Hemer
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Universitätsklinikum Münster, Münster
  - Mathias-Spital Rheine, Rheine
- Greece (7):
  - "Hippokratio" Hospital of Athens, 2nd Internal Medicine Clin, Athens
  - General Hospital of Chest Diseases Sotiria, Athens
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Larisa, Oncology Clinic, Larissa
  - General Hospital of Larissa, Larissa
  - Metropolitan Hospital, Oncology Clinic, Neo Faliro, Athens
  - General Hospital "G. Papageorgiou", Thessaloniki
- Hungary (9):
  - National Koranyi TBC and Pulm. Internal Med. Clinic, Budapest
  - Semmelweis University, Budapest
  - Institute of Chest Diseases Csongrad County,Dpt. Pulmonology, Deszk
  - Pulmonology Institute of Veszprem County, Farkasgyepu, Farkasgyepü
  - Aladar Petz County Teaching Hospital, Dept. Pulmonology, Győr
  - Lung Hospital of Matra, Dept. Pulmonology, Mátraháza
  - Josa Andras Korhaz, Nyiregyhaza, Nyíregyháza
  - University of Pecs, 1st internal Med. Dept., Pulmonology, Pécs
  - Pest County Lung Hospital, Department No. 3, Törökbálint
- India (8):
  - Vikram Hospital, Bangalore
  - V S Hospital, Chennai
  - Dr. Kamakshi Memorial Hospital, Chennai
  - Sri Ramachandra Medical College & Research Institute, Chennai
  - M.S. Patel Cancer Hospital, Karamsad
  - B. P .Poddar Hospital & Medical Research Ltd., Kolkata, West Bengal
  - Tata Memorial Hospital, Mumbai
  - Ruby Hall Clinic, Pune
- St James's Hospital, Dublin, Ireland
- Italy (11):
  - P.O. Bellaria IRCCS Istituto delle scienze Neurologiche di Bologna, Bologna
  - ASST di Cremona, Cremona
  - Spedali Riuniti di Livorno, Livorno
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera di Parma, Parma
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Ospedale San Vincenzo, Taormina (ME)
  - Ospedale Molinette, AO Città della Salute e della, Torino
  - A. O. S. Maria della Misericordia, Udine
- Mexico (3):
  - Instituto Nacional de Cancerologia, México
  - Hospital y Clínica OCA S. A. de C. V., Monterrey
  - Centro Hemato-Oncologico Privado de Toluca S.A. de C.V., Toluca
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis-Hertogenbosch, 's-Hertogenbosch
  - Rijnstate Hospital, Arnhem
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - METC Academisch Ziekenhuis Maastricht/Universiteit van Maastricht, Maastricht
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- Portugal (6):
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - CHLN, EPE - Hospital de Santa Maria, Lisbon
  - IPO Lisboa Francisco Gentil, EPE, Lisbon
  - IPO Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar São João,EPE, Porto
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Singapore (2):
  - National Cancer Centre, Singapore
  - Johns Hopkins Singapore International Medical Centre, Singapore
- South Korea (9):
  - Chungbuk National University Hospital, Cheongju-si
  - Gachon University Gil Medical Center, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - The Catholic University of Korea, St.Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
- Spain (9):
  - Hospital A Coruña, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clínico de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Taiwan (9):
  - Chang Gung Memorial Hospital Chiayi, Chiayi City
  - Buddhist Tzu Chi General Hospital, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yet-Sen Cancer Center, Taipei
  - Taipe Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital(TaoYuan), Taoyuan District
- Turkey (Türkiye) (8):
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Uludag Universitesi Tip Fakultesi, Bursa, Bursa
  - Dicle Universitesi Tip Fakultesi, Diyarbakır
  - Gaziantep Univ. Tip Fakultesi Tibbi Onkoloji Bilim Dali, Gaziantep
  - Kartal Egitim Ve Arastirma Hastanesi, Istanbul
  - Yedikule Gog. Hst. EAH, Istanbul
  - Ege Universitesi Tip Fakultesi Tibbi Onkoloji Bilim Dali, Izmir
  - Dr.Suat Seren EAH, Izmir
- United Kingdom (10):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Harrogate District Hospital, Harrogate
  - Royal Free Hospital, London
  - The Royal Marsden Hospital, London
  - Maidstone Hospital, Kent Oncology Centre, Maidstone
  - Nottingham City Hospital, Nottingham
  - Scarborough Hospital, Scarborough
  - The Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Lu S, Li W, Zhou C, Hu CP, Qin S, Cheng G, Feng J, Wang J, Cseh A, Peil B, Gibson N, Ehrnrooth E, Zhang L. Afatinib vs erlotinib for second-line treatment of Chinese patients with advanced squamous cell carcinoma of the lung. Onco Targets Ther. 2018 Nov 30;11:8565-8573. doi: 10.2147/OTT.S161506. eCollection 2018. PMID 30573970
- [Derived] Goss GD, Felip E, Cobo M, Lu S, Syrigos K, Lee KH, Goker E, Georgoulias V, Li W, Guclu S, Isla D, Min YJ, Morabito A, Ardizzoni A, Gadgeel SM, Fulop A, Buhnemann C, Gibson N, Kramer N, Solca F, Cseh A, Ehrnrooth E, Soria JC. Association of ERBB Mutations With Clinical Outcomes of Afatinib- or Erlotinib-Treated Patients With Lung Squamous Cell Carcinoma: Secondary Analysis of the LUX-Lung 8 Randomized Clinical Trial. JAMA Oncol. 2018 Sep 1;4(9):1189-1197. doi: 10.1001/jamaoncol.2018.0775. PMID 29902295
- [Derived] Gadgeel S, Goss G, Soria JC, Felip E, Georgoulias V, Lu S, Cobo M, Syrigos K, Lee KH, Goker E, Guclu SZ, Isla D, Morabito A, Dupuis N, Buhnemann C, Kramer N, Solca F, Ehrnrooth E, Ardizzoni A. Evaluation of the VeriStrat(R) serum protein test in patients with advanced squamous cell carcinoma of the lung treated with second-line afatinib or erlotinib in the phase III LUX-Lung 8 study. Lung Cancer. 2017 Jul;109:101-108. doi: 10.1016/j.lungcan.2017.05.010. Epub 2017 May 11. PMID 28577938
- [Derived] Soria JC, Felip E, Cobo M, Lu S, Syrigos K, Lee KH, Goker E, Georgoulias V, Li W, Isla D, Guclu SZ, Morabito A, Min YJ, Ardizzoni A, Gadgeel SM, Wang B, Chand VK, Goss GD; LUX-Lung 8 Investigators. Afatinib versus erlotinib as second-line treatment of patients with advanced squamous cell carcinoma of the lung (LUX-Lung 8): an open-label randomised controlled phase 3 trial. Lancet Oncol. 2015 Aug;16(8):897-907. doi: 10.1016/S1470-2045(15)00006-6. Epub 2015 Jul 5. PMID 26156651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-Label Phase-III trial to compare the efficacy of afatinib with erlotinib for the second-line treatment of patients with advanced non-small cell lung cancer, who completed at least 4 cycles of platinum-based doublet chemotherapy. Randomization ratio was 1:1. Stratification was based on race.
Pre-assignment Details: Patients screened to ensure that they met all inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria were not met. Tumor assessments at screening were completed within 21 days and other screening assessments were completed within 28 days, of randomization.
Groups:
- Afatinib: Patients administered 40 milligram (mg) film-coated tablet once daily orally for the first 28-day treatment course. Dose escalation to 50 mg once daily was allowed at the beginning of the second 28-day treatment course, if patients met specified safety and compliance criteria. Dose reduction to 40 mg/day (if applicable), 30 mg/day, or 20 mg/day, was required in the presence of known drug-related adverse events.
- Erlotinib: Patients administered 150 mg film-coated tablet once daily orally, with dose reduction to 100 mg/day or 50 mg/day in the presence of known drug-related adverse events.
Period: Overall Study
Arm/Group | Afatinib | Erlotinib
Started | 398 | 397
Treated | 392 | 395
Completed | 0 | 0
Not Completed | 398 | 397
Not completed — Other than listed | 5 | 5
Not completed — Worsening of underlying cancer disease | 19 | 34
Not completed — Adverse Event | 68 | 52
Not completed — Protocol Violation | 5 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 28 | 20
Not completed — Withdrew due to Progressive disease | 265 | 279
Not completed — Randomised but bot treated | 6 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Set (RS): All patients who were randomized, regardless of whether they received investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib | Erlotinib | Total
Number analyzed (Participants) | 398 | 397 | 795
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Randomised set
  Years | 64.9 (8.39) | 63.4 (8.98) | 64.1 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Randomised set
  Participants
    Female | 63 | 66 | 129
    Male | 335 | 331 | 666
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not captured in this trial. Population: Randomised set
  Participants
    American Indian or Alaska Native | 2 | 2 | 4
    Asian | 97 | 94 | 191
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 7 | 8 | 15
    White | 288 | 291 | 579
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival, Based on Central Independent Review as Determined by Response Evaluation Criteria in Solid Tumours 1.1
Description: Progression Free Survival (PFS) was defined as the time from randomization to disease progression (or death if the patient died before progression) by central independent review according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. RECIST is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize") or worsen ("progress") during treatment. Per RECIST v1.1 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: First treatment administration up until cut off date of 02 March 2015 (up to 1058 days).
Population: Randomized Set (RS): All patients who were randomized, regardless of whether they received investigational treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib | Erlotinib
Number analyzed (Participants) | 398 | 397
Months | 2.63 [2.00 to 2.86] | 1.94 [1.87 to 2.10]
Statistical Analysis 1: Comparison: Afatinib vs Erlotinib; A Cox proportional hazards model without the randomization stratification variable was used for each subgroup category, along with the corresponding log-rank test; Test type: Superiority or Other; p = 0.0103, Log Rank — P-value from log-rank stratified by Race (two-sided). Hazard ratio (Afatinib vs Erlotinib) from Cox proportional hazards model stratified by Race; Hazard Ratio (HR) = 0.814, 95% CI 2-sided [0.693 to 0.956]

2. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from randomisation to death. It was a key secondary endpoint.
Time Frame: From first drug administration from 9 April 2012 until study closure on 27 Dec 2017 (approximately 2089 days).
Population: RS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib | Erlotinib
Number analyzed (Participants) | 398 | 397
Months | 7.82 [7.19 to 8.71] | 6.77 [5.85 to 7.79]
Statistical Analysis 1: Comparison: Afatinib vs Erlotinib; A Cox proportional-hazards model, stratified by race, was used to estimate the hazard ratio and 95% confidence interval (CI) between the two treatment groups; Test type: Superiority or Other; p = 0.0193, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.841, 95% CI 2-sided [0.727 to 0.973]

3. Secondary Outcome: Number of Participants With Objective Response According to RECIST 1.1
Description: A patient with a best overall response of Complete Responder (CR) or Partial Responder (PR) was considered to show objective response to study medication. For patients with an objective response, time to objective response was defined as the time from randomization to the first objective response; duration of objective response was defined as the time from the first objective response to progression (or death if the patient died before progression). Per RECIST v1.1 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: First treatment administration up until cut off date of 02 March 2015 (up to 1058 days).
Population: RS
Measure: Number; unit: Participants
Arm/Group | Afatinib | Erlotinib
Number analyzed (Participants) | 398 | 397
Participants | 22 | 11
Statistical Analysis 1: Comparison: Afatinib vs Erlotinib; Test type: Superiority or Other; p = 0.0551, Regression, Logistic — Odds ratio (Afatinib vs Erlotinib), 95% CI and p-value (two-sided) from logistic regression stratified by race; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.98 to 4.32]

4. Secondary Outcome: Number of Participants With Disease Control According to RECIST 1.1
Description: Disease control was assessed based on Independent Radiologic Review (IRR) and investigator assessment. A patient with a best overall response of CR, PR, or Stable Disease (SD) was considered to have disease control. Patients with no baseline target lesions who had no evidence of disease progression in their non-target lesions and had no new lesions were considered to have disease control. Per RECIST v1.1 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: First treatment administration up until cut off date of 02 March 2015 (up to 1058 days).
Population: RS
Measure: Number; unit: Participants
Arm/Group | Afatinib | Erlotinib
Number analyzed (Participants) | 398 | 397
Participants | 201 | 157
Statistical Analysis 1: Comparison: Afatinib vs Erlotinib; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds ratio (Afatinib vs Erlotinib), 95% CI and p-value (two-sided) from logistic regression stratified by race; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.18 to 2.06]

5. Secondary Outcome: Tumour Shrinkage
Description: Maximum percentage decrease from baseline in the sum of target lesion diameters following independent review. The change in the size (i.e. the sum of diameters (SOD)) of target lesions from baseline was derived. Tumour shrinkage for each patient was measured (based on Independent Radiologic Review (IRR)) as the minimum SOD of target lesions after randomisation.
  A negative percentage indicates decrease from baseline; positive numbers indicate an increase of tumour size. The mean maximum decrease from baseline of +5 and +9.4 reflect an average increase in tumour size.
  Post-baseline mean is adjusted for baseline sum of diameters and race.
Time Frame: First treatment administration up until cut off date of 02 March 2015 (up to 1058 days).
Population: Patients from the randomised set with tumour assessments are considered for the analysis of this endpoint.
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | Afatinib | Erlotinib
Number analyzed (Participants) | 307 | 311
Millimeter (mm) | 78.8 (1.26) | 80.0 (1.24)
Statistical Analysis 1: Comparison: Afatinib vs Erlotinib; The analysis will compare the treatments using analysis of covariance (ANCOVA) for minimum sum of diameters, using baseline sum of diameters as a covariate. The randomization strata will be included as classification factors; Test type: Superiority or Other; p = 0.500, ANCOVA; Adjusted mean = -1.2, 95% CI 2-sided [-4.67 to 2.28], Standard Error of Mean 1.77 — Mean was adjusted for baseline sum of diameters and race

6. Secondary Outcome: Number of Participants With Status Change in Cough, Dyspnoea and Pain Related Items Over Time in Health Related Quality of Life Questionnaire
Description: Health-related quality of life (HRQoL) was measured with the following multi-dimensional questionnaires: the european organization for research and treatment of cancer (eortc) quality of life questionnaire (QLQ-C30) questionnaire and its lung cancer specific supplementary module EORTC QLQ-LC13 and the EQ-5D health status self-assessment questionnaire. The questionnaires were assessed at the first visit of each treatment course, at end of treatment (EOT) and follow up prior to clinical assessment. The results displayed show number of patients with improvement in the relevant criteria. For each of the summary scales and items measuring cough, dyspnoea and pain, the two treatment arms were compared in terms of: The number of patients that were improved: Change in cough; dyspnoea and pain scores over time.
Time Frame: From first drug administration from 9 April 2012 until study closure on 27 Dec 2017 (approximately 2089 days).
Population: RS
Measure: Number; unit: Participants
Arm/Group | Afatinib | Erlotinib
Number analyzed (Participants) | 398 | 397
Participants
  Improved Cough: number analyzed (Participants) | 339 | 341
  Improved Cough | 147 | 120
  Improved Dyspnoea: number analyzed (Participants) | 339 | 340
  Improved Dyspnoea | 174 | 150
  Improved Pain Related: number analyzed (Participants) | 343 | 342
  Improved Pain Related | 138 | 134
  Improved Global Health Status: number analyzed (Participants) | 339 | 339
  Improved Global Health Status | 121 | 96

7. Secondary Outcome: Summary of Time to Deterioration in Coughing, Dyspnoea and Pain.
Description: Health-related quality of life (HRQoL) was measured with the following multi-dimensional questionnaires: the EORTC QLQ-C30. The questionnaires were assessed at the first visit of each treatment course. For each of the summary scales and items measuring cough, dyspnoea and pain, the two treatment arms were compared in terms of: Time to deterioration.
Time Frame: From first drug administration from 9 April 2012 until study closure on 27 Dec 2017 (approximately 2089 days).
Population: RS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib | Erlotinib
Number analyzed (Participants) | 398 | 397
Months
  Time to Deterioration - Coughing: number analyzed (Participants) | 180 | 182
  Time to Deterioration - Coughing | 4.53 [2.86 to 4.93] | 3.65 [2.79 to 4.66]
  Time to Deterioration - Dyspnoea: number analyzed (Participants) | 238 | 244
  Time to Deterioration - Dyspnoea | 2.63 [1.97 to 2.86] | 1.91 [1.87 to 2.33]
  Time to Deterioration - Pain: number analyzed (Participants) | 243 | 232
  Time to Deterioration - Pain | 2.50 [2.00 to 2.79] | 2.37 [1.91 to 2.76]
Statistical Analysis 1: Comparison: Afatinib vs Erlotinib; The results shown relate to Time to Deterioration in Coughing; Test type: Superiority or Other; p = 0.2562, Regression, Cox — p-value calculated using log rank test stratified by race; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.72 to 1.09] — Hazard ratio (Afatinib vs Erlotinib) from Cox proportional hazard model stratified by race
Statistical Analysis 2: Comparison: Afatinib vs Erlotinib; The results shown relate to Time to Deterioration in Dyspnoea; Test type: Superiority or Other; p = 0.0078, Regression, Cox — p-value calculated using log rank test stratified by race; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.66 to 0.94] — Hazard ratio (Afatinib vs Erlotinib) from Cox proportional hazard model stratified by race
Statistical Analysis 3: Comparison: Afatinib vs Erlotinib; The results shown relate to Time to Deterioration in Pain; Test type: Superiority or Other; p = 0.8690, Regression, Cox — p-value calculated using log rank test stratified by race; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.82 to 1.18] — Hazard ratio (Afatinib vs Erlotinib) from Cox proportional hazard model stratified by race

8. Secondary Outcome: Change in Score Over Time in Coughing,Dyspnoea and Pain
Description: Health related quality of life (HRQoL) was measured with the following multi dimensional questionnaires: the EORTC QLQ-C30. The questionnaires were assessed at the first visit of each treatment course. For each of the summary scales and items measuring cough, dyspnoea and pain, the two treatment arms were compared in terms of change in score over time, adjusted for baseline score and race.
  Questionnaires have items relating to Cough, Dyspnoea and Pain. Overall Scores are transformed to a standardised scale of 0 to 100 with the larger value indicating a worse outcome. A change of (+/-) 10 points is considered to be relevant.
  The change in cough, dyspnea and pain will be assessed using a mixed effects growth curve model with the average profile over time for each endpoint described by a piecewise linear model (presented as post baseline in data table). Post-baseline mean is adjusted for baseline and race.
Time Frame: From first drug administration from 9 April 2012 until study closure on 27 Dec 2017 (approximately 2089 days).
Population: RS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Afatinib | Erlotinib
Number analyzed (Participants) | 398 | 397
Units on a scale
  Coughing: number analyzed (Participants) | 340 | 333
  Coughing | 15.8 (2.40) | 19.3 (2.37)
  Dyspnoea: number analyzed (Participants) | 340 | 332
  Dyspnoea | 11.4 (1.83) | 14.9 (1.85)
  Pain: number analyzed (Participants) | 343 | 334
  Pain | 10.3 (2.13) | 13.1 (2.17)
Statistical Analysis 1: Comparison: Afatinib vs Erlotinib; The results shown relate to Change in scores over time for: Coughing; Test type: Superiority or Other; p = 0.0091, Regression, Cox; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-6.15 to -0.88], Standard Error of Mean 1.34
Statistical Analysis 2: Comparison: Afatinib vs Erlotinib; The results shown relate to Change in scores over time for: Dyspnoea; Test type: Superiority or Other; p = 0.0024, Regression, Cox; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-5.75 to -1.25], Standard Error of Mean 1.15
Statistical Analysis 3: Comparison: Afatinib vs Erlotinib; The results shown relate to Change in scores over time for: Pain; Test type: Superiority or Other; p = 0.0384, Regression, Cox; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-5.33 to -0.15], Standard Error of Mean 1.32

ADVERSE EVENTS:
Time Frame: From first drug administration from 9 April 2012 until study closure on 27 Dec 2017 (approximately 2089 days).
Description: All adverse events (AEs) reported for this trial are on treatment AEs.
Arm/Group | Afatinib | Erlotinib
All-Cause Mortality (participants affected / at risk) | 77/392 | 71/395
Serious Adverse Events (participants affected / at risk) | 174/392 | 175/395
Other Adverse Events (participants affected / at risk) | 383/392 | 371/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=392) | Erlotinib (N=395)
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 2
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 4
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2
Pericarditis (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0
Aphagia (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 18 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 3
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 1
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5
Asthenia (General disorders) | 6 | 3
Chest discomfort (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 6
Condition aggravated (General disorders) | 1 | 1
Death (General disorders) | 4 | 2
Device occlusion (General disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 11 | 6
Mucosal inflammation (General disorders) | 2 | 1
Multi-organ failure (General disorders) | 1 | 1
Necrosis (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 2 | 3
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 4
Sudden death (General disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 6
Bronchopneumonia (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 2 | 5
Oral fungal infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 26 | 16
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 9 | 2
Septic shock (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Blood calcium increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 1
Blood urea increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 12 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 | 16
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 3 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 2 | 4
Dysarthria (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2
Motor dysfunction (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 2
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1
Bladder mass (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 9 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 30
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 12
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Haemorrhage (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 1
Inferior vena cava syndrome (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=392) | Erlotinib (N=395)
Anaemia (Blood and lymphatic system disorders) | 31 | 41
Constipation (Gastrointestinal disorders) | 43 | 42
Diarrhoea (Gastrointestinal disorders) | 284 | 158
Nausea (Gastrointestinal disorders) | 81 | 62
Stomatitis (Gastrointestinal disorders) | 54 | 21
Vomiting (Gastrointestinal disorders) | 48 | 38
Asthenia (General disorders) | 61 | 48
Chest pain (General disorders) | 14 | 20
Fatigue (General disorders) | 65 | 67
Mucosal inflammation (General disorders) | 50 | 14
Pyrexia (General disorders) | 32 | 33
Paronychia (Infections and infestations) | 41 | 18
Weight decreased (Investigations) | 38 | 51
Decreased appetite (Metabolism and nutrition disorders) | 94 | 100
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 25
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 23
Dizziness (Nervous system disorders) | 12 | 21
Insomnia (Psychiatric disorders) | 20 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 65 | 67
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 68 | 69
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 44 | 39
Productive cough (Respiratory, thoracic and mediastinal disorders) | 14 | 21
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 38 | 56
Dry skin (Skin and subcutaneous tissue disorders) | 36 | 47
Pruritus (Skin and subcutaneous tissue disorders) | 38 | 52
Rash (Skin and subcutaneous tissue disorders) | 196 | 187

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT01523587/Prot_000.pdf
  • Statistical Analysis Plan (2012-04-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT01523587/SAP_001.pdf